CLINICAL TRIAL: NCT06295783
Title: Prospective Evaluation of the Relation Between Different Questionnaires Measuring Radiation-induced Side-effect
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1059; NCI-2024-01955 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Cancer (HNC) Questionnaire: Participants will be asked to fill out three head and neck cancer (HNC) questionnaires during your visits to the clinic:
  1. The MDASI-HN questionnaire (standard-of-care) has 28 questions.
  2. The EORTC QLQ-HN35 questionnaire has 35 questions.
  3. The EORTC QLQ-30 questionnaire has 30 questions.
  Interventions: Other: MDASI-HN; Other: EORTC QLQ-C30; Other: EORTC HN35

INTERVENTIONS:
Other: MDASI-HN — Given by Questionnaire
Other: EORTC QLQ-C30 — Given by Questionnaire
Other: EORTC HN35 — Given by Questionnaire

SUMMARY:
To learn more about how you would rate the intensity or severity of your symptoms during or after radiation therapy using questionnaires with different rating scales.

DETAILED DESCRIPTION:
Primary Objectives:

• To investigate how different toxicity questionnaires with different scoring systems can be reliably translated to each other by estimating different measures of correlation between items and summary scores across different questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* English as a primary language
* Participants with a diagnosis of HNC undergoing active curative RT or having received curative RT within the past 5 years at MD Anderson
* Ability to complete the survey(s) of their own volition

Exclusion Criteria:

* Age < 18 years
* Non-English speaking participants
* Participants who are receiving or have received RT in a non-HN site.
* Participants in follow up and over 5 years from post-treatment
* Neurocognitive deficits that render patients unable to complete the survey(s) on their own.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and Neck Cancer (HNC) participants undergoing active radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Moreno, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org